CLINICAL TRIAL: NCT06242548
Title: How Type I Diabetes Responds to Different Diets (Normoglucidic or Ketogenic) During Physical Activity at Altitude
Acronym: DIAREAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHMS23001
Record Dates: First submitted 2023-04-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-06

CONDITIONS: Diet Habit; Type I Diabetes; Activity, Motor; Control
Keywords: type I diabetes; diet (normoglucidic or ketogenic); physical activity at altitude
MeSH Terms: conditions — Feeding Behavior; Diabetes Mellitus, Type 1; Motor Activity | interventions — Blood Glucose; Weights and Measures; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: a group of type 1 diabetes patients and to a group of controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- physical activity at altitude while maintaining usual diet (Other): organisation of physical activity outings in the mountains at a level already practised by the subjects, while maintaining their usual diet (normoglucidic or ketogenic); '.
  collection of capillary blood samples (blood sugar, ketone levels), non-invasive biometric data (weight, oxygen saturation by transcutaneous sensor), and questionnaires (BORG scale, food consumption before/during/after exercise).
  Interventions: Other: physical activity outings in the mountains at a level already practised by the subjects, while maintaining their usual diet (normoglucidic or ketogenic)

INTERVENTIONS:
Other: physical activity outings in the mountains at a level already practised by the subjects, while maintaining their usual diet (normoglucidic or ketogenic) — organisation of 4 physical activity outings in the mountains at a level already practised by the subjects, while maintaining their usual diet (normoglucidic or ketogenic).
  During each of of the 4 physical activity outings, collection of capillary blood samples (blood sugar, ketone levels), non-invasive biometric data (weight, oxygen saturation by transcutaneous sensor), and questionnaires (BORG scale, food consumption before/during/after exercise).
  Other Names: collection of capillary blood samples (blood sugar, ketone levels); collection of non-invasive biometric data (weight, oxygen saturation by transcutaneous sensor); questionnaires (BORG scale, food consumption before/during/after exercise)

SUMMARY:
To date, no study has shown the effects of diets (normoglucidic or ketogenic) on type I diabetes during physical activity (hiking, ski touring) at altitude.

The ketogenic diet in the general population is increasingly studied scientifically, but no clinical trial has studied it in type I diabetic patients during physical activity at altitude. Similarly, no study has investigated the effects of this diet on ketone and blood glucose levels in athletes during physical activity at altitude.

Therefore, its impact on blood glucose and ketone levels during exercise at altitude is unknown in healthy and type I diabetic subjects.

Since the investigators are studying ketonemia at altitude, and since ketonemia depends on insulin and carbohydrate intake, it is necessary to also study a control group with the same diet, in order to analyse whether the results obtained at altitude are related to the diet alone or to the diet in the context of diabetes.

In order to avoid certain biases and confounding factors, the type I diabetic group will be compared to a control group of healthy subjects, in which the subjects have the same diet as the diabetic group.

This is a pioneering study, of significant interest because the ketogenic diet is recent and rapidly increasing in interest in diabetic patients, with no scientific data for mountain physical activity. Doctors, diabetologists and sports doctors, are still without data to advise their diabetic patients who wish to follow a ketogenic diet on the benefits/risks of this diet, or to explain to them how to react to physical activity in the mountains.

DETAILED DESCRIPTION:
To date, no study has shown the effects of diets (normoglucidic or ketogenic) on type I diabetes during physical activity (hiking, ski touring) at altitude.

Today, many sportsmen and women use the ketogenic diet (reproducing the effects of food fasting) because it improves physical performance. In particular, it avoids the undesirable effects of carbohydrate intake during re-sugaring (digestive level, fatigue, glycaemic peak) and reduces muscular fatigue.

Patients with type II diabetes also use this diet because insulin resistance decreases, weight loss is increased, and diabetes is balanced.

The ketogenic diet in the general population is increasingly studied scientifically, but no clinical trial has studied it in type I diabetic patients during physical activity at altitude. Similarly, no study has investigated the effects of this diet on ketone and blood glucose levels in athletes during physical activity at altitude.

Therefore, its impact on blood glucose and ketone levels during exercise at altitude is unknown in healthy and type I diabetic subjects.

Since the investigators are studying ketonemia at altitude, and since ketonemia depends on insulin and carbohydrate intake, it is necessary to also study a control group on the same diet, in order to analyse whether the results obtained at altitude are related to the diet alone or to the diet in the context of diabetes.

In order to avoid certain biases and confounding factors, the type I diabetic group will be compared to a control group of healthy subjects, in which the subjects have the same diet as the diabetic group.

This is a pioneering study, of significant interest because the ketogenic diet is recent and rapidly increasing in interest in diabetic patients, with no scientific data for mountain physical activity. Doctors, diabetologists and sports doctors, are still without data to advise their diabetic patients who wish to follow a ketogenic diet on the benefits/risks of this diet, or to explain to them how to react to physical activity in the mountains.

The main objective is the effect of normoglucidic and ketogenic diets on diabetic parameters (blood glucose and ketone levels) during physical activity at altitude in type I diabetics in comparison with the control group.

The secondary objective is to evaluate the effect of diets (normoglucidic or ketogenic) on physical skills during a physical activity (hiking, ski touring) at a peak altitude during the outing at 2000m and 2500m in both groups.

Each participant must agree to take part in 2 mountain physical activity outings at 2000m and 2 outings at 2500m. The physical activity must be similar in nature (hiking or skiing) and pace.

All outings are supervised (by the Diamachro association and the co-investigator for the diabetes group and by the co-investigator for the control group).

the sequence of the 4 outings will be the same, including blood glucose and ketone measurements, heart rate and oxygen saturation measurements, as well as the completion by the subject of the food collection and the Borg scale.

After the data have been collected, they will be analysed by the investigator

ELIGIBILITY:
Inclusion Criteria:

For the diabetes group:

* Major subjects with type I diabetes, enrolled in the Diamachro association in conjunction with the diabetology department of the Centre Hospitalier Métropole Savoie in Chambéry
* treated with insulin in basal/bolus form or on pump
* regularly (>2x/month) doing physical activity (hiking or ski touring) at altitude (>1500m)
* agreeing to make 4 mountain outings (hiking or ski touring): 2 at an altitude of 2000m and 2 at an altitude of 2500m
* be affiliated to, or benefit from, a health insurance scheme.

For the control group:

* major subjects with no known endocrine pathology.
* Regularly (>2x/month) engaged in physical activity (hiking or ski touring) at altitude (>1500m)
* agreeing to do 4 mountain outings (hiking or ski touring): 2 at an altitude of 2000m and 2 at an altitude of 2500m
* be affiliated to, or benefit from, a health insurance scheme.
* healthy adults who usually go out in the mountains

Exclusion Criteria:

For the diabetes group:

* minor subject
* subject with diabetes other than type I diabetes
* adult under guardianship, curatorship, or judicial protection

For the control group:

* minor subject
* adult under guardianship, trusteeship, or court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Glycemia variation among groups over time during mountains outings | each hours from one hour before the start of the outing to one hours after the start of the outing. Each outing will last 8 hours.
  The primary outcome will be the variation of glycemia (mmol/l - capillary blood sampling) among groups over outing's time assessed using a linear mixed effect model including as fixed effect the outing effect (n=4), the time effect (cf. Time frame) and the group effect (+/- diabetes) and as random effect the subject number. This model will allow the test of the group:time interaction effect with a control of the outings effect (replicate condition) to match the primary outcome.
Ketonemia variation among groups over time during mountains outings | each hours from one hour before the start of the outing to one hours after the start of the outing. Each outing will last 8 hours.
  The primary outcome will be the variation of ketonemia (mmol/l - capillary blood sampling) among groups over outing's time assessed using a linear mixed effect model including as fixed effect the outing effect (n=4), the time effect (cf. Time frame) and the group effect (+/- diabetes) and as random effect the subject number. This model will allow the test of the group:time interaction effect with a control of the outings effect (replicate condition) to match the primary outcome.

SECONDARY OUTCOMES:
heart rate variation among groups over time during mountains outings | each hours from one hour before the start of the outing to one hours after the start of the outing. Each outing will last 8 hours.
  This secondary outcome will be the variation of heart rate (bpm - heart rate monitor) among groups over outing's time assessed using a linear mixed effect model including as fixed effect the outing effect (n=4), the time effect (cf. Time frame) and the group effect (+/- diabetes) and as random effect the subject number. This model will allow the test of the group:time interaction effect with a control of the outings effect (replicate condition) to match this secondary outcome.
oxygen saturation variation among groups over time during mountains outings | each hours from one hour before the start of the outing to one hours after the start of the outing. Each outing will last 8 hours.
  This secondary outcome will be the variation of oxygen saturation (% - pulse oxymeter) among groups over outing's time assessed using a linear mixed effect model including as fixed effect the outing effect (n=4), the time effect (cf. Time frame) and the group effect (+/- diabetes) and as random effect the subject number. This model will allow the test of the group:time interaction effect with a control of the outings effect (replicate condition) to match this secondary outcome.
Evaluation of physical skills assessment during each of the 4 mountains outings | at the end of the outing (8 hours from the start)
  evaluation by the subject, by completing the Borg scale; 1= no effort (better outcome). 10=maximal effort (worse outcome)
assessment of food intake for each of the 4 mountains outings | 24h before the outings and at the end of the outing (8 hours from the start)
  amount of food ingested in grams, reported by the subject in a food diary
weight measurements for each of the 4 mountains outings | 12h before the outings and at the end of the outing (8 hours from the start)
  measurement of the weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Moulin, Principal Investigator — Centre Hospitalier Métropole Savoie
Locations (1):
- Marie-Christine Carret, Chambéry, Cente Hospitalier Métropole Savoie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehair S. Intérêt des régimes hypoglucidiques pour la prise en charge du diabète : revue de la littérature. Thèse presented at; 2018 Feb 22.
- [Result] Fu S, Li L, Deng S, Zan L, Liu Z. Effectiveness of advanced carbohydrate counting in type 1 diabetes mellitus: a systematic review and meta-analysis. Sci Rep. 2016 Nov 14;6:37067. doi: 10.1038/srep37067. PMID 27841330
- [Result] Feinman RD, Pogozelski WK, Astrup A, Bernstein RK, Fine EJ, Westman EC, Accurso A, Frassetto L, Gower BA, McFarlane SI, Nielsen JV, Krarup T, Saslow L, Roth KS, Vernon MC, Volek JS, Wilshire GB, Dahlqvist A, Sundberg R, Childers A, Morrison K, Manninen AH, Dashti HM, Wood RJ, Wortman J, Worm N. Dietary carbohydrate restriction as the first approach in diabetes management: critical review and evidence base. Nutrition. 2015 Jan;31(1):1-13. doi: 10.1016/j.nut.2014.06.011. Epub 2014 Jul 16. PMID 25287761
- [Result] Harcombe Z, Baker JS, DiNicolantonio JJ, Grace F, Davies B. Evidence from randomised controlled trials does not support current dietary fat guidelines: a systematic review and meta-analysis. Open Heart. 2016 Aug 8;3(2):e000409. doi: 10.1136/openhrt-2016-000409. eCollection 2016. PMID 27547428
- [Result] Riddell MC, Gallen IW, Smart CE, Taplin CE, Adolfsson P, Lumb AN, Kowalski A, Rabasa-Lhoret R, McCrimmon RJ, Hume C, Annan F, Fournier PA, Graham C, Bode B, Galassetti P, Jones TW, Millan IS, Heise T, Peters AL, Petz A, Laffel LM. Exercise management in type 1 diabetes: a consensus statement. Lancet Diabetes Endocrinol. 2017 May;5(5):377-390. doi: 10.1016/S2213-8587(17)30014-1. Epub 2017 Jan 24. PMID 28126459
- [Result] de Mol P, de Vries ST, de Koning EJ, Gans RO, Tack CJ, Bilo HJ. Increased insulin requirements during exercise at very high altitude in type 1 diabetes. Diabetes Care. 2011 Mar;34(3):591-5. doi: 10.2337/dc10-2015. Epub 2011 Jan 27. PMID 21273491
- [Result] Matejko B, Gawrecki A, Wrobel M, Hohendorff J, Benbenek-Klupa T, Zozulinska-Ziolkiewicz D, Malecki MT, Klupa T. Physiological Characteristics of Type 1 Diabetes Patients during High Mountain Trekking. J Diabetes Res. 2020 Sep 15;2020:8068710. doi: 10.1155/2020/8068710. eCollection 2020. PMID 33015195
- [Result] Malcolm G, Rilstone S, Sivasubramaniyam S, Jairam C, Chew S, Oliver N, Hill NE. Managing diabetes at high altitude: personal experience with support from a Multidisciplinary Physical Activity and Diabetes Clinic. BMJ Open Sport Exerc Med. 2017 Aug 16;3(1):e000238. doi: 10.1136/bmjsem-2017-000238. eCollection 2017. PMID 29021909
- [Result] Zajac A, Poprzecki S, Maszczyk A, Czuba M, Michalczyk M, Zydek G. The effects of a ketogenic diet on exercise metabolism and physical performance in off-road cyclists. Nutrients. 2014 Jun 27;6(7):2493-508. doi: 10.3390/nu6072493. PMID 24979615
- [Result] Langfort J, Pilis W, Zarzeczny R, Nazar K, Kaciuba-Uscilko H. Effect of low-carbohydrate-ketogenic diet on metabolic and hormonal responses to graded exercise in men. J Physiol Pharmacol. 1996 Jun;47(2):361-71. PMID 8807563